CLINICAL TRIAL: NCT02158338
Title: Do Bonding Disruptions Occur More Often in Children With Asthma Than in Non-asthmatic Populations?
Status: Completed | Type: Observational
Sponsor: Ran Anbar (Other)
Responsible Party: Sponsor-Investigator, Ran Anbar, Professor, State University of New York - Upstate Medical University
Organization: State University of New York - Upstate Medical University (Other)
Other Study IDs: 389127
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Asthma in Children; Anxiety
Keywords: asthma; maternal bonding; maternal bonding disruptions; mother-infant interaction
MeSH Terms: conditions — Anxiety Disorders; Asthma | interventions — NPSR1 protein, human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asthma: Mothers of children thought to have asthma
  Interventions: Other: Asthma
- Non-asthma: Mothers of children without diagnosed respiratory problems
  Interventions: Other: Non-asthma

INTERVENTIONS:
Other: Asthma — mothers who have children that have been diagnosed with respiratory issues
  Groups: Asthma
Other: Non-asthma — mothers who have children that do not have a diagnosis of respiratory problems
  Groups: Non-asthma

SUMMARY:
Six studies have preceded this project. Three studies suggested that there is a significant connection between pediatric asthma and disruptions in maternal-infant bonding (Feinberg, 1988; Schwartz, 1988; Pennington, 1991). Three studies suggested that children with asthma benefit from a type of therapy that improves bonding with their mothers (Madrid, Ames, Skolek, & Brown, 2000; Madrid, Ames, Horner, Brown, & Navarrette, 2004; Madrid, Pennington, Brown & Wolfe, 2011).

This study proposes to study in a more thorough fashion the question of the incidence of bonding disruptions with between mothers and their children with asthma. This time there will be a larger sample, and more stringent criteria will used in assigning children to the asthma cohort. Through questions answered by mothers whose children have been said to have asthma, we will be able to decide if the children's respiratory conditions are likely to be attributable to asthma or more likely reflective of another respiratory condition such as vocal cord dysfunction or anxiety related hyperventilation (Anbar, 2014).

ELIGIBILITY:
Inclusion Criteria:

* Biological mothers of male and female children between 2 and 12 years of age who live with or have contact with their children
* English is the primary language of the biological mother

Exclusion Criteria:

* Mothers of children only below 2 or above 12 years of age
* Mothers of children thought to have a chronic health condition other than asthma
* Mothers who have already completed a questionnaire with another child

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with asthma and/or maternal infant bonding issues | Day 1
  A questionnaire will be scored by a pediatric pulmonologist and a psychologist

CONTACTS AND LOCATIONS:
Overall Officials: Ran D Anbar, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Background] Anbar, R.D. Functional symptoms in pulmonology: taking your breath away. In: Ran D. Anbar (ed), Functional Symptoms in Pediatric Disease: A Clinical Guide. New York, NY: Springer, 2014; 47-58.
- [Background] Anbar RD, Geisler SC. Identification of children who may benefit from self-hypnosis at a pediatric pulmonary center. BMC Pediatr. 2005 Apr 25;5(1):6. doi: 10.1186/1471-2431-5-6. PMID 15850484
- [Background] Annesi-Maesano I, Moreau D, Strachan D. In utero and perinatal complications preceding asthma. Allergy. 2001 Jun;56(6):491-7. doi: 10.1034/j.1398-9995.2001.056006491.x. PMID 11421892
- [Background] Feinberg, Steven. Degree of maternal infant bonding and its relationship to pediatric asthma and family environments. Unpublished doctoral dissertation, Professional School of Psychology, San Francisco, 1988.
- [Background] Kero J, Gissler M, Gronlund MM, Kero P, Koskinen P, Hemminki E, Isolauri E. Mode of delivery and asthma -- is there a connection? Pediatr Res. 2002 Jul;52(1):6-11. doi: 10.1203/00006450-200207000-00004. PMID 12084840
- [Background] Klaus, M. H., & Kennen, J. H. Maternal-infant bonding. St. Louis, MO: C. V. Mosby, 1976.
- [Background] Klinnert MD, Nelson HS, Price MR, Adinoff AD, Leung DY, Mrazek DA. Onset and persistence of childhood asthma: predictors from infancy. Pediatrics. 2001 Oct;108(4):E69. doi: 10.1542/peds.108.4.e69. PMID 11581477
- [Background] Kozyrskyj AL, Mai XM, McGrath P, Hayglass KT, Becker AB, Macneil B. Continued exposure to maternal distress in early life is associated with an increased risk of childhood asthma. Am J Respir Crit Care Med. 2008 Jan 15;177(2):142-7. doi: 10.1164/rccm.200703-381OC. Epub 2007 Oct 11. PMID 17932381
- [Background] Madrid A. Helping children with asthma by repairing maternal-infant bonding problems. Am J Clin Hypn. 2005 Oct-2006 Jan;48(2-3):199-211. doi: 10.1080/00029157.2005.10401517. PMID 16482847
- [Background] Mantymaa M, Puura K, Luoma I, Salmelin R, Davis H, Tsiantis J, Ispanovic-Radojkovic V, Paradisiotou A, Tamminen T. Infant-mother interaction as a predictor of child's chronic health problems. Child Care Health Dev. 2003 May;29(3):181-91. doi: 10.1046/j.1365-2214.2003.00330.x. PMID 12752609
- [Background] Nafstad P, Samuelsen SO, Irgens LM, Bjerkedal T. Pregnancy complications and the risk of asthma among Norwegians born between 1967 and 1993. Eur J Epidemiol. 2003;18(8):755-61. doi: 10.1023/a:1025395405101. PMID 12974550
- [Background] Pennington, D. Events associated with maternal-infant bonding deficits and severity of pediatric asthma. Unpublished doctoral dissertation, Professional School of Psychology, San Francisco, 1991.
- [Background] Schwartz, M.P. Incidence of events associated with maternal-infant bonding disturbance in a pediatric population. Unpublished doctoral dissertation, Rosebridge Graduate School, Walnut Creek, 1988.
- [Background] Roduit C, Scholtens S, de Jongste JC, Wijga AH, Gerritsen J, Postma DS, Brunekreef B, Hoekstra MO, Aalberse R, Smit HA. Asthma at 8 years of age in children born by caesarean section. Thorax. 2009 Feb;64(2):107-13. doi: 10.1136/thx.2008.100875. Epub 2008 Dec 3. PMID 19052046
- [Background] Wright RJ, Cohen S, Carey V, Weiss ST, Gold DR. Parental stress as a predictor of wheezing in infancy: a prospective birth-cohort study. Am J Respir Crit Care Med. 2002 Feb 1;165(3):358-65. doi: 10.1164/ajrccm.165.3.2102016. PMID 11818321
- [Background] Wright RJ, Visness CM, Calatroni A, Grayson MH, Gold DR, Sandel MT, Lee-Parritz A, Wood RA, Kattan M, Bloomberg GR, Burger M, Togias A, Witter FR, Sperling RS, Sadovsky Y, Gern JE. Prenatal maternal stress and cord blood innate and adaptive cytokine responses in an inner-city cohort. Am J Respir Crit Care Med. 2010 Jul 1;182(1):25-33. doi: 10.1164/rccm.200904-0637OC. Epub 2010 Mar 1. PMID 20194818